CLINICAL TRIAL: NCT02423122
Title: A Clinical Study of Two Doses of a Selective p38 MAP Kinase Inhibitor, VX-745, to Evaluate the Effects of 12-Week Oral Twice-Daily Dosing on Amyloid Plaque Load as Assessed by Quantitative Dynamic 11C-PiB Positive Emission Tomography (PET) Amyloid Scanning
Brief Title: A PET Study of the Effects of p38 MAP Kinase Inhibitor, VX-745, on Amyloid Plaque Load in Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP-VX00-745-302
Record Dates: First submitted 2015-04-14; First posted 2015-04-22 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — VX-745

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX-745 dose 1 (Experimental): Active Group 1: VX-745 40 mg twice daily
  Interventions: Drug: VX-745
- VX-745 dose 2 (Experimental): Active Group 2: VX-745 125 mg twice daily
  Interventions: Drug: VX-745

INTERVENTIONS:
Drug: VX-745 — Orally-Active Selective P45 MAP Kinase inhibitor

SUMMARY:
This study will assess the effects of administration of VX-745 for 12 weeks on amyloid plaque burden in Alzheimer's disease (AD). Subjects who meet entry criteria will undergo 11C-PiB (Carbon-11-labeled Pittsburgh Compound B) positron emission tomography (PET) at baseline and after 45 days of dosing with VX-745. Cognitive testing will also be conducted at baseline and day 45.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Diagnosis of mild cognitive impairment (MCI) due to probable AD or of mild AD
* MMSE range: 20 to 28
* Evidence of amyloid pathology by amyloid PET scan
* Participants may be taking medications for AD, provided that the dose of these medications has been stable for >3 months
* Proficiency in Dutch and adequate visual and auditory abilities to be able to perform all aspects of the cognitive and functional tests
* Adequate visual and auditory abilities to perform all aspects of the cognitive and functional assessments.

Exclusion Criteria:

* Evidence of neurodegenerative disease other than AD
* Inability for any reason to undergo PET and fMRI scans (including notably: history of allergic reaction of any severity to 11C-PiB injection; pacemaker, vascular stent or stent graft)
* Psychiatric disorder that would compromise ability to comply with study requirements
* Significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder or metabolic/endocrine disorders or other disease that would preclude treatment with p38 MAP kinase inhibitor and/or assessment of drug safety and efficacy
* Recent (<90 days) changes to AD medications prescribed for cognitive reasons or with the potential to impact cognition
* Participation in a study of an investigational drug less than 6 months or 5 half-lives of the investigational drug, whichever is longer, before enrollment in the study
* Male subjects with female partner of child-bearing potential who are unwilling or unable to adhere to contraception requirements
* Female subjects who have not reached menopause or have not had a hysterectomy or bilateral oophorectomy/salpingoophorectomy
* Positive urine or serum pregnancy test or plans desires to become pregnant during the course of the trial
* Any factor deemed by the investigator to be likely to interfere with study conduction

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Scheltens, MD, Principal Investigator — Alheimer Research Center, VU medisch centrum
Locations (1):
- Alzheimer Research Center, VU Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Tormahlen NM, Martorelli M, Kuhn A, Maier F, Guezguez J, Burnet M, Albrecht W, Laufer SA, Koch P. Design and Synthesis of Highly Selective Brain Penetrant p38alpha Mitogen-Activated Protein Kinase Inhibitors. J Med Chem. 2022 Jan 27;65(2):1225-1242. doi: 10.1021/acs.jmedchem.0c01773. Epub 2021 May 11. PMID 33974419

RESULTS

PARTICIPANT FLOW:
Groups:
- Neflamapimod (VX-745) Dose 1: Active Group 1: VX-745 40 mg twice daily
  VX-745: Orally-Active Selective P45 MAP Kinase inhibitor
- Neflamapimod (VX-745) Dose 2: Active Group 2: VX-745 125 mg twice daily
  VX-745: Orally-Active Selective P45 MAP Kinase inhibitor
Period: Overall Study
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2 | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 76] | 65 [60 to 75] | 66.5 [60 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Amyloid Plaque Burden by 11C-PiB PET
Description: Percent change in global cortical amyloid specific PET signal (BPND)
Time Frame: Baseline compared to following 12 weeks' dosing with VX-745
Population: All patients with baseline and Day 84 11C-PiB scan. One patient in 40 mg dose group could not cooperate for Day 84 PET scan due to having developed MRI-induced panic attack.
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2
Number analyzed (Participants) | 8 | 7
percentage change from baseline | -4.57 [-11.65 to 4.83] | 4.57 [0.56 to 12.25]

2. Primary Outcome: Number of 11C-PiB Responders
Description: Number of patients meeting protocol pre-specified definition of response: > 7% reduction in global cortical BPND
Time Frame: Day 84
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2
Number analyzed (Participants) | 8 | 7
Participants | 3 | 1

3. Secondary Outcome: Wechsler Memory Scale (WMS) Immediate Recall Composite
Description: WMS immediate-recall composite score consisted of the sum of the scores on Logical Memory I, Verbal Paired Associates I, and Visual Reproduction I. The composite score ranges from 0 to 136; with higher score indicating better performance.
Time Frame: Baseline to Day 84
Population: All patients with baseline and day 84 WMS testing data. One subject in 40 mg dose group did not complete the Day 84 WMS assessment after having developed MRI-induced panic attack.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2
Number analyzed (Participants) | 8 | 7
units on a scale | 7.0 (11.0) | 13.4 (12.2)

4. Secondary Outcome: Wechsler Memory Scale (WMS) Delayed Recall Composite
Description: WMS delayed-recall composite score at each testing sessions consisted of the sum of the scores on Logical Memory II, Verbal Paired Associates II, and Visual Reproduction II. The composite score ranges from 0 to 136; with higher scores indicating better performance.
Time Frame: Change from baseline to Day 84
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neflamapimod (VX-745) Dose 1 | Neflamapimod (VX-745) Dose 2
Number analyzed (Participants) | 8 | 7
units on a scale | 7.5 (7.0) | 10.4 (11.9)

ADVERSE EVENTS:
Arm/Group | 40 mg Dose Group | 125 mg Dose Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 6/9 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg Dose Group (N=9) | 125 mg Dose Group (N=7)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less